CLINICAL TRIAL: NCT03488576
Title: Macular Peeling With Foveal Sparing of the Internal Limiting Membrane: A Pilot Study
Brief Title: Foveal Sparing of the ILM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Francesco Semeraro, Francesco Semeraro; MD, Associate Professor, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitreo003
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Retinal Sensitivity

STUDY DESIGN:
Intervention Model Description: This was a prospective study including ninety-one eyes of 190 phakic patients scheduled to undergo vitrectomy for idiopathic macular pucker or macular hole, from July 2014 to December 2016. Patients were randomized in a 1:1 ratio to complete peeling of the ILM (CP group) or foveal sparing (FS group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete Peeling (Active Comparator): Patient underwent scheduled vitrectomy for epiretinal membrane or macular hole with complete macular peeling of the internal limiting membrane.
  Interventions: Procedure: Complete Macular Peeling
- Foveal Sparing (Experimental): Patient underwent scheduled vitrectomy for epiretinal membrane or macular hole with partial peeling the internal limiting membrane (foveal sparing).
  Interventions: Procedure: Macular Peeling with Foveal Sparing

INTERVENTIONS:
Procedure: Complete Macular Peeling — A complete peeling of the internal limiting membrane was performed
  Arms: Complete Peeling
Procedure: Macular Peeling with Foveal Sparing — A partial peeling of the internal limiting membrane was performed, sparing the fovea.
  Arms: Foveal Sparing

SUMMARY:
To compare the retinal sensitivity of complete internal limiting membrane (ILM) peeling versus foveal sparing ILM peeling during vitrectomy for epiretinal membrane or macular hole.

ELIGIBILITY:
Inclusion Criteria:

* provision of written informed consent
* age > 60 years
* presence of idiopathic macular pucker or macular hole documented by OCT

Exclusion Criteria:

* any prior intraocular surgery
* pathologic myopia (> 7 diopters)
* age related macular degeneration
* glaucoma and diabetic retinopathy or any other retinal vascular disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Retinal Sensitivity (dB) | 12-month
  Microperimetry was done to assess macular sensitivity
Visual Acuity (LogMAR) | 12-month
  ETDRS charts were used to assess best corrected visual acuity
Central Retinal Thickness (microns) | 12-month
  Optical Coherence Tomography will be used to assess central retinal thickness

IPD SHARING:
Plan to Share IPD: No